CLINICAL TRIAL: NCT05022875
Title: Effectiveness of the 'Healthcare CEO' App for Type 1 Diabetes Patients Transitioning From Adolescence to Early Adulthood: Protocol for a Randomized Controlled Trial
Brief Title: Effectiveness of The Health Care CEO App for T1D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yueh-Tao Chiang, Assistant Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ChangGungUCEOApp
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; transition; mobile health; treatment fidelity
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Experimental group: The complete Healthcare chief executive officer app will be used for intervention in the experimental group.
  Control Group: Participants in the control group will only install the "CEO's Profile" and "Health Tracking" interfaces of the Healthcare chief executive officer app.
Who Masked: Participant, Care Provider
Masking Description: Blinding strategies include the following: (1) the statistician will not be allowed to disclose the randomization results to others; (2) after physician referral, the participant will be immediately ushered to a separate room to ensure that the caregiver does not receive information regarding the intervention content; and (3) participants of both the experimental and control groups will download the app, but app content will be different between the two groups. (4) research assistants will specially emphasize for all participants that app usage is beneficial for disease management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental app intervention (Experimental): The complete Healthcare CEO app will be used for intervention in the experimental group.
  Interventions: Device: Healthcare CEO app- for experimental app intervention
- Control app intervention (Sham Comparator): Participants in the control group will only install the "CEO's Profile" and "Health Tracking" interfaces of the Healthcare CEO app.
  Interventions: Device: Healthcare CEO app-for control app intervention

INTERVENTIONS:
Device: Healthcare CEO app- for experimental app intervention — The app content was designed based on the results of previous qualitative and Delphi studies (Chiang et al., 2021; Chiang et al., 2020) and consists of 11 interfaces: CEO's profile, Health Tracking, CEO Knowledge Base, Barrier-free Communication, See Here: Diet and Exercise, Help Me, Detective!, CEO Chatroom, CEO's Secretary, Who's the Best CEO, SOS Calls, and Q&A
  Arms: Experimental app intervention
Device: Healthcare CEO app-for control app intervention — consists of 2 interfaces: CEO's profile, Health Tracking.
  Arms: Control app intervention

SUMMARY:
The present study aims to evaluate the intervention effectiveness of the Healthcare Chief Executive Officer mobile application(Healthcare CEO app) in patients with type 1 diabetes transitioning from adolescence to early adulthood.

DETAILED DESCRIPTION:
Aim:The present study aims to evaluate the intervention effectiveness of the Healthcare Chief Executive Officer mobile application in patients with type 1 diabetes transitioning from adolescence to early adulthood.

Design: A 9-month two-arm, parallel-group, single-blind, randomized controlled trial Methods: Ninety-six Type-1 diabetes patients, aged 16-25 years, are expected to participate in this study. Participants will be randomly assigned to the experimental or control group by central randomization. The Healthcare Chief Executive Officer app, which consists of the following functions: data recording, knowledge, communication skills, food swap guide, exercise recommendations, chatroom, reminders, and SOS, will be used as the intervention measure. We will compare the differences in disease control outcomes, confidence in self-management, self-care behaviors, emotional distress, quality of life, and specific diabetes-related knowledge between the two groups before intervention and at 3, 6, and, 9 months post-intervention. The differences within the experimental group pre- and post- intervention will also be analyzed. This study design was approved by the ethics committee of the researcher's affiliation in March 2021.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of T1D by an endocrinologist before the age of 16 and a disease duration of >6months
* patients aged 16-25 years
* mean HbA1C level ≥7.5% one year before inclusion
* ability to communicate in Chinese or Mandarin
* patients who own smartphones with internet access
* patients who agreed to voice recording during a session explaining the treatment process
* patients who signed the informed consent form prior to participation; for minors, a legal representative must provide consent and sign the informed consent form.

Exclusion Criteria:

･ T1D patients with other concomitant metabolic diseases, chromosomal aberrations, major illnesses, and cognitive impairment will be excluded from this study.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline and 3, 6, 9 months
  HbA1c from baseline to 9months
Change in % with HbA1c <7.0% | Baseline and 3, 6, 9 months
  Percentage of individuals in each group with HbA1c <7.0%
Change in Hyperglycemic Events | Baseline and 3, 6, 9 months
  Number of events of each participant with blood sugar >200 mg/dl or" high" on glucometer, Ketoacidosis diagnosed
Change in Hypoglycemic Events | Baseline and 3, 6, 9 months
  Number of events of each participant with blood sugar <60 mg/dl or "low" on glucometer, Hypoglycemia diagnosed

SECONDARY OUTCOMES:
Change in Perceived Diabetes Self-Management Scale score over time | Baseline and 3, 6, 9 months
  Perceived Diabetes Self-Management Scale (PDSMS):The original questionnaire was developed by Wallston et al. (2007). It consists of 8 items scored on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree),The translated questionnaire has content validity, Cronbach's α, and test-retest reliability values of 0.75, 0.93, and 0.97, respectively.
Change in Self-care Behavior Assessment Scale score over time | Baseline and 3, 6, 9 months
  Self-care Behavior Assessment Scale: This scale was developed by Wang (2010) to measure self-care behaviors of adolescents with T1D. A total of 39 items are scored on a 5-point Likert scale ranging from 1 (not achieved at all) to 5 (completely achieved). The total score ranges from 39 to 195, with higher scores indicating better self-care behaviors. Cronbach's α and the content validity index (CVI) value based on content rating by experts are 0.87 and 0.92, respectively.
Change in Diabetes Distress Scale score over time | Baseline and 3, 6, 9 months
  Diabetes Distress Scale (DDS): The original scale was developed by Polonsky et al. (2005). The Chinese version consists of 18 items across four subscales. Items are scored on a 4-point Likert scale ranging from 1 (no distress) to 4 (severely distressed), with higher scores indicating more severe emotional distress. Cronbach's α and test-retest reliability values of the DDS were 0.89 and 0.81, respectively (Liu et al., 2010).
Change in Diabetes Quality of Life Scale score over time | Baseline and 3, 6, 9 months
  Diabetes Quality of Life (DQOL): The original scale was developed for use in the Diabetes Control and Complications Trial and was translated in Chinese by Cheng et al. (1999).Higher scores are indicative of higher QOL. Cronbach's α and test-retest reliability values of the scale and subscales are within the ranges of 0.76-0.92 and 0.94-0.99, respectively.
Change in Diabetes Knowledge Questionnaire score over time | Baseline and 3, 6, 9 months
  Diabetes Knowledge Questionnaire (DKQ): The original questionnaire was developed by Garcia et al. (2001). The Chinese version comprises 24 items that are answered "Yes," "No" or "I don't know"; 1 point is awarded for each correct answer. The total score ranges from 0 to 24 points.reliability and Cronbach's α values of 0.78 and 0.89, respectively (Hu et al., 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Tao Chiang, PhD, Study Director — Chang Gung University; Fu-Sung Lo, BSN, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang-Gung University and Chang-Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chiang YT, Yu HY, Tsay PK, Chen CW, Chang CW, Hsu CL, Lo FS, Moons P. Effectiveness of the User-Centered "Healthcare CEO" App for Patients With Type 1 Diabetes Transitioning From Adolescence to Early Adulthood: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 13;14:e59871. doi: 10.2196/59871. PMID 39805107